CLINICAL TRIAL: NCT04695496
Title: The Application of Repetitive Transcranial Magnetic Stimulation on the Freezing of Gait in People With Parkinson's Disease
Brief Title: Repetitive Transcranial Magnetic Stimulation on Freezing of Gait in People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chien Tai Hong, Doctorate of Medicine and of Philosophy, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202003057
Record Dates: First submitted 2020-11-22; First posted 2021-01-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theta bust stimulating group (Experimental): Theta burst stimulation with Magstim super rapid 2, over SMA. 3 section per day, for 5 days, total 15 sections.
  Interventions: Device: Theta bust stimulating

INTERVENTIONS:
Device: Theta bust stimulating — Theta burst stimulation with Magstim super rapid 2, over SMA. 3 section per day, for 5 days, total 15 sections.

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease. The cardinal symptoms of PD are tremor, rigidity, bradykinesia and postural instability. Gait disturbance is also one of the key features of PD. At present, the mainstream treatment of PD is the dopaminergic supplement. However, the response to the medical treatment varies between symptoms. Rigidity and bradykinesia respond to the medical treatment the best, and tremor respond partially. Gait disorders do not usually respond to the dopaminergic medication. Freezing of gait (FOG) is one of the most notorious and devastating presentation of gait disorders in PD. Currently, there is no available treatment for FOG, even the invasive deep brain stimulation does not work on it. Repetitive transcortical magnetic stimulation (rTMS) is a novel non-invasive intervention. Through the magnetic stimulation, brain neurons could be activated by the electrical current. The application of rTMS had been approved by US FDA for the treatment of depression. The possible effect of rTMS may result from the stimulation-related neuronal plasticity. Regarding PD, rTMS also had been found to had some effect on different motor symptoms, mainly on the bradykinesia and rigidity but not gait. The present study would like to test the accumulative effect of rTMS on gait disorders of PD, especially the phenomenon of FOG. All the study subjects will receive rTMS under intermittent theta burst stimulation (iTBS) mode at supplementary motor area (SMA). Gait analysis and other motor performance will be assessed before and after the intervention.

DETAILED DESCRIPTION:
The present trial is designed as an open-label, uncontrolled pilot study for evaluating the effect of rTMS on improvement of freezing of gait (FOG) in people with PD. The primary endpoint is the improvement of FOG, and the secondary endpoint is the improvement of motor symptoms and cognition. All participants need to complete the informed consent before they are enrolled into the trial. Demographic data includes age, sex, medical history, drug history, disease duration, modified Hoehn-Yahr stage, and UPDRS score are collected. Gait function are evaluated with time up and go (TUG), freezing of gait questionnaire (FOG-Q), and Gait-up device analysis before trial starting. Cognitive function including mini-mental state examination (MMSE), clocking drawing test, Wechsler memory scale (WMS)-world list test and spatial span test, trial making test A and B, category fluency test (animal naming), and beck depression inventory-II are tested by trained neuropsychiatrists. Pre-treatment brain image examined by magnetic resonance image (MRI) and blood sampling for synapse protein level are performed. The participants are then arranged to receive theta burst stimulation for 5 days by Magstim Rapid® system (Super Rapid 2) equipped with air cooled coil (D70), stimulating on supplementary motor area (SMA). After the intervention, post-treatment evaluation including gait function, motor symptoms, cognition, brain MRI, and blood sampling will be performed again with the same methods at 1 month later. Any adverse event during the trial period will also be recorded. The trial is expected to be conducted in Shuang-Ho hospital, Taipei Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease, age between 45-80 years old.
2. Can walk independently for 10 meters
3. With FOG at either on or off period of time

Exclusion Criteria:

- People with

1. pre-existing and active major neurological diseases other than PD
2. with a previous history of seizures
3. with implanted metallic objects that would contraindicate rTMS
4. unable to perform fMRI
5. with skin damage on the stimulation area
6. with multiple sclerosis
7. with large ischemic scars
8. with a family history or medical history of seizures, epilepsy
9. brain damage may affect the threshold for inducing epilepsy
10. taken tricyclic antidepressants, analgesics, or anything that may lower the threshold for inducing epilepsy
11. with sleep disorders during the rTMS treatment
12. with severe alcohol abuse or use of epilepsy drugs
13. with severe heart disease or uncontrollable migraine caused by high intracranial pressure
14. who are actively suicidal during the trial period, have recurring major medical disorders, or with neurological co-morbidities such as space occupying lesions, CVA, aneurysms etc

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of duration on time up an go (TUG) test at 1 months later after theta burst stimulation | Baseline and 1 months later after theta burst stimulation
  Measurement change of duration on time up an go (TUG) test
Change of score on freezing of gait questionnaire (FOG-Q) at 1 months later after theta burst stimulation | Baseline and 1 months later after theta burst stimulation
  Measurement change of score on freezing of gait questionnaire (FOG-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Tai Hong, MD, PHD, Study Chair — Shuang Ho hospital, Taipei Medical University
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Some of participants hesitate to share their IPD.